CLINICAL TRIAL: NCT02257346
Title: The Effect of Perioperative Systemic Lidocaine on Quality of Recovery After Cesarean Delivery
Brief Title: Intravenous Lidocaine and Quality of Recovery After Cesarean Delivery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI terminated study with no subjects enrolled.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jason Farrer, Clinical Instructor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Lidocaine-RCT
Record Dates: First submitted 2014-07-16; First posted 2014-10-06 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy
Keywords: Pregnancy; Lidocaine; Quality; Recovery
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Intravenous lidocaine 1.5 mg/Kg bolus dose and 2mg/Kg/hr infusion
  Interventions: Drug: Lidocaine
- Normal Saline (Placebo Comparator): Intravenous normal saline infusion
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine — Lidocaine infusion will be administered immediately after delivery of the fetus and continue through 1 hour into recovery period.
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Normal Saline — Normal Saline will be administered as a placebo immediately after delivery of the fetus and continue through 1 hour into recovery period
  Other Names: 0.9% Saline
  Arms: Normal Saline

SUMMARY:
When given intravenously, the local anesthetic lidocaine has been shown to decrease the amount of pain medication patients require when recovering from several types of surgeries. Cesarean delivery is a very common surgery in the United States, effecting more than 1 million women each year. The investigators hypothesize that lidocaine, given during and immediately after a patient undergoes a cesarean section, will help improve a mother's overall recovery experience, as well as positively influence bonding with her new baby.

DETAILED DESCRIPTION:
Pain after Cesarean delivery is a common occurrence on the labor and delivery unit. The increased use of neuraxial anesthesia has allowed the administration of neuraxial opioids to help with postoperative pain control. Many patients, however, still require IV and oral opioids in the post anesthesia recovery unit (PACU), and on the postpartum nursing floor. Post Cesarean delivery pain not only has the usual adverse effects common to all postoperative pain (i.e. increased risk for deep vein thrombosis, pulmonary embolism, coronary ischemia, pneumonia, poor wound healing, and psychological dysfunction) but also has the potential to adversely affect mother-baby bonding, time spent in skin-to-skin contact and success of initiating effective breastfeeding.

Systemic administration of lidocaine has been shown to decrease opioid consumption, improve recovery of bowel function and promote a better recovery after inpatient procedures. Lidocaine has been shown to have analgesic, antihyperalgesic and anti-inflammatory properties. It also has an excellent safety profile when given by a low-dose infusion.

Assessing a patient's quality of recovery has become an important outcome in several studies. The patient's capacity to return to her normal activities and effectively care for her newborn is one of the most important signs of a successful surgical procedure, and it has significant economic, sociological and psychological implications.

Quality of recovery -40(QoR-40) is a validated 40-item instrument to assess the quality of post-operative recovery (10). Myles et al. have concluded that the QoR-40 would be a useful outcome measure to assess the impact on changes in health care delivery, but anesthesia studies underutilize this instrument.

This study will evaluate the effect of perioperative systemic lidocaine in the postoperative quality of recovery of patients undergoing Cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Class II
* English speaking
* Scheduled Cesarean delivery

Exclusion Criteria:

* Allergy to local anesthetics
* Chronic opioid use
* Greater than 2 prior cesarean deliveries
* Prior myomectomy
* Prior classical cesarean incision
* BMI greater than 40
* History of cardiac disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2015-02-15 (Actual); Study Completion 2015-02-15 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 40 on the day after surgery | 1 day
  The quality of recovery 40 (QoR-40) is a validated questionnaire used to assess several variables that effect a patient's post-operative experience.

SECONDARY OUTCOMES:
Opioid consumption | 1 day
  Total opioid consumption for the first 24 hours after delivery
Skin-to-skin time | 1 day
  Percentage of time a patient spends in skin to skin contact with their newborn in the first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Farrer, M.D., Principal Investigator — Northwestern University
Locations (1):
- NorthwesternUniversity, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bramson L, Lee JW, Moore E, Montgomery S, Neish C, Bahjri K, Melcher CL. Effect of early skin-to-skin mother--infant contact during the first 3 hours following birth on exclusive breastfeeding during the maternity hospital stay. J Hum Lact. 2010 May;26(2):130-7. doi: 10.1177/0890334409355779. Epub 2010 Jan 28. PMID 20110561
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Gill TM, Feinstein AR. A critical appraisal of the quality of quality-of-life measurements. JAMA. 1994 Aug 24-31;272(8):619-26. PMID 7726894
- [Background] Guyatt GH, Cook DJ. Health status, quality of life, and the individual. JAMA. 1994 Aug 24-31;272(8):630-1. No abstract available. PMID 8057520
- [Background] Watcha MF, Issioui T, Klein KW, White PF. Costs and effectiveness of rofecoxib, celecoxib, and acetaminophen for preventing pain after ambulatory otolaryngologic surgery. Anesth Analg. 2003 Apr;96(4):987-994. doi: 10.1213/01.ANE.0000053255.93270.31. PMID 12651647
- [Background] Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, Nagy A, Rubinstein A, Ponsford JL. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesth Analg. 1999 Jan;88(1):83-90. doi: 10.1097/00000539-199901000-00016. PMID 9895071
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540